### **CLINICAL STUDY PROTOCOL**

IND - 145417

# An Open-Label, Multicenter Study to Evaluate the Safety and Efficacy of Repeat Intramuscular ABP-450 (prabotulinumtoxinA) Injection for the Treatment of Cervical Dystonia

### **ABP-19002**

| Sponsor: | Aeon Biopharma, Inc. |
|---|---|
| <b>Sponsor Contact:</b> | |
| Medical Monitor: | |
| Version of Protocol: | Version 2.1 |
| Date of Protocol: | 13 May 2021 |
| | 18 March 2020 (Version 1.0)<br>26 August 2020 (Version 1.1) |
| | 03 December 2020 (Version 2.0) |

#### CONFIDENTIAL

All financial and non-financial support for this study will be provided by Aeon Biopharma, Inc. The concepts and information contained in this document or generated during the study are considered proprietary and may not be disclosed in whole or in part without the expressed, written consent of Aeon Biopharma, Inc.

The study will be conducted according to the International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) guideline E6 (R2): Good Clinical Practice (GCP).

# Protocol Approval - Sponsor Signatory

**Study Title** 

An Open-Label, Multicenter Study to Evaluate the Safety and Efficacy

of Repeat Intramuscular ABP-450 (prabotulinumtoxinA) Injection for

the Treatment of Cervical Dystonia

Protocol Number

ABP-19002

**Protocol Date** 

13 May 2021; Version 2.1

and Version

Protocol accepted and approved by:

Vice President, Technical Operations and Regulatory

Signature

Date Date

# Protocol Approval – Principal/Coordinating Investigator

Study Title An Open-Label, Multicenter Study to Evaluate the Safety and Efficacy

of Repeat Intramuscular ABP-450 (prabotulinumtoxinA) Injection for

the Treatment of Cervical Dystonia

Protocol Number ABP-19002

**Protocol Date** 

13 May 2021; Version 2.1

and Version

Protocol accepted and approved by:

Principal/Coordinating Investigator

Sign 5/17/2021

## Protocol Approval - Principal/Coordinating Investigator

**Study Title** 

An Open-Label, Multicenter Study to Evaluate the Safety and Efficacy

of Repeat Intramuscular ABP-450 (prabotulinumtoxinA) Injection for

the Treatment of Cervical Dystonia

Protocol Number

ABP-19002

**Protocol Date** 

13 May 2021; Version 2.1

and Version

Protocol accepted and approved by:

### Principal/Coordinating Investigator

| | 5/17/21 |
|-----------|---------|
| Signature | Date |

## Protocol Approval - Lead Statistician

| Study Title | An Open-Label, | Multicenter Study to | Evaluate the Safety and |
|---|---|---|---|
|---|---|---|---|

Efficacy of Repeat Intramuscular ABP-450 (prabotulinumtoxinA)

Injection for the Treatment of Cervical Dystonia

Protocol Number ABP-19002

**Protocol Date** 13 May 2021; Version 2.1

and Version

Protocol accepted and approved by:

Lead Statistician

Signature Date

## Protocol Approval - Medical Monitor

Study Title An Open-Label, Multicenter Study to Evaluate the Safety and

Efficacy of Repeat Intramuscular ABP-450 (prabotulinumtoxinA)

Injection for the Treatment of Cervical Dystonia

Protocol Number ABP-19002

Protocol Date 13 1

13 May 2021; Version 2.1

and Version

Protocol accepted and approved by:

#### **Medical Monitor**



### **Declaration of Investigator**

I have read and understood all sections of the protocol entitled "An Open-Label, Multicenter Study to Evaluate the Safety and Efficacy of Repeat Intramuscular ABP-450 (prabotulinumtoxinA) Injection for the Treatment of Cervical Dystonia" and the accompanying investigator's brochure.

I agree to supervise all aspects of the protocol and to conduct the clinical investigation in accordance with the Final Protocol Version 2.1, dated 13 May 2021, the International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) guideline E6 (R2): Good Clinical Practice (GCP) and all applicable government regulations. I will not make changes to the protocol before consulting with Aeon Biopharma, Inc. or implement protocol changes without independent ethics committee approval except to eliminate an immediate risk to patients. I agree to administer investigational study drug only to patients under my personal supervision or the supervision of a subinvestigator.

I will not supply the investigational drug to any person not authorized to receive it. Confidentiality will be protected. Patient identity will not be disclosed to third parties or appear in any study reports or publications.

I will not disclose information regarding this clinical investigation or publish results of the investigation without authorization from Aeon Biopharma, Inc.

| Signature of Principal Investigator | Date |
|----------------------------------------|----------|
| | <u>_</u> |
| Printed Name of Principal Investigator | |

# **Table of Contents**

| Tab | le of ( | Contents | | 8 |
|---|---|---|---|---|
| List | of Ta | ıbles | | 11 |
| Pro | tocol | Synopsis | 5 | 12 |
| List | of Al | bbreviati | ons | 22 |
| 1 | Intro | duction. | | 24 |
| 2 | Stud | y Object | ives and Estimands | 27 |
| | 2.1 | - | Objectives | |
| | | 2.1.1 | Primary Objective | |
| | | 2.1.2 | Secondary Objective | |
| | 2.2 | Study I | Estimands | |
| | | 2.2.1 | Target Population | 27 |
| | | 2.2.2 | Primary Estimand | |
| | | 2.2.3 | Secondary Estimands | 28 |
| 3 | Inve | stigation | al Plan | 29 |
| | 3.1 | Study I | Design | 29 |
| | | 3.1.1 | Rationale of Study Design | 29 |
| | | 3.1.2 | Conduct of the Study During the COVID-19 Pandemic | |
| 4 | Patie | ent Selec | tion and Withdrawal Criteria | 31 |
| | 4.1 | Selection | on of Study Population | 31 |
| | | 4.1.1 | Inclusion Criteria | 31 |
| | | 4.1.2 | Exclusion Criteria | 32 |
| | | 4.1.3 | Rescreening. | 33 |
| | 4.2 | Withdra | awal of Patients from the Study | 33 |
| | | 4.2.1 | Reasons for Withdrawal/Discontinuation | 33 |
| | | 4.2.2 | Handling of Withdrawals | 34 |
| | | 4.2.3 | Replacements | |
| 5 | Stud | y Treatm | nents | 35 |
| | 5.1 | Method | d of Assigning Patients to Treatment Group | 35 |
| | 5.2 | Treatment Administered | | 35 |
| | 5.3 | Identity | of Investigational Product | 37 |

| | 5.4 | Manage | ement of Clinical Supplies | 37 |
|---|---|---|---|---|
| | | 5.4.1 | Investigational Study Drug Packaging and Storage | 37 |
| | | 5.4.2 | Test Article Accountability | |
| | | 5.4.3 | Other Supplies. | |
| | 5.5 | Overdos | se Management | 38 |
| | | 5.5.1 | Treatment of Overdose | 38 |
| | 5.6 | Blinding | g | 38 |
| | | 5.6.1 | Breaking the Blind | 38 |
| | 5.7 | Treatme | ent Compliance | |
| | 5.8 | Prior an | d Concomitant Therapy | 39 |
| 6 | Stud | y Assessr | nents and Procedures | 40 |
| | 6.1 | Study V | isits | 40 |
| | 6.2 | Safety A | Assessments | 42 |
| | | 6.2.1 | Adverse Events | 43 |
| | | 6.2.1.1 | Definitions of Adverse Events | 43 |
| | | 6.2.1.2 | Serious Adverse Events | 43 |
| | | 6.2.1.3 | Eliciting and Documenting Adverse Events | 43 |
| | | 6.2.1.4 | Reporting Adverse Events | 44 |
| | | 6.2.1.5 | Reporting Serious Adverse Events | 45 |
| | | 6.2.1.6 | Suspected Unexpected Serious Adverse Reactions and Non-Serious Adverse Events of Special Interest | 45 |
| | | 6.2.1.7 | Assessment of Severity | 46 |
| | | 6.2.1.8 | Assessment of Causality | 46 |
| | | 6.2.1.9 | Follow-Up of Patients Reporting Adverse Events | 47 |
| | 6.3 | Seconda | ary Efficacy Assessments | 48 |
| | | 6.3.1 | TWSTRS Scale | 48 |
| | | 6.3.2 | PGI-C and CGI-C Scales | 49 |
| | | 6.3.4 | C-SSRS | 49 |
| | | 6.3.5 | Dysphagia Score | |
| | 6.4 | | Monitoring Committee | |
| | J | ~~100, 1 | | |

| | | harma, Inc.<br>BP-19002 (Version 2.1) | ABP-450<br>13 May 2021 |
|---|---|---|---|
| | 6.5 | Pregnancy | 50 |
| | 6.6 | Laboratory Analyses | 50 |
| | 6.7 | Sample Collections | 51 |
| 7 | Statis | stical Considerations | 52 |
| | 7.1 | Estimands | 52 |
| | 7.2 | Sample Size Calculations | 52 |
| | 7.3 | Analysis Sets | 52 |
| | 7.4 | Description of Subgroups to be Analyzed | 53 |
| | 7.5 | Statistical Analysis Methodology | 53 |
| | | 7.5.1 Analysis of Primary Estimand | 53 |
| | | 7.5.2 Analysis of Secondary Estimands | 53 |
| | | 7.5.3 Other Analyses | 54 |
| | | 7.5.4 Interim Analyses | 54 |
| 8 | Data | Quality Assurance | 55 |
| | 8.1 | Data Management | 55 |
| 9 | Ethic | es | 56 |
| | 9.1 | Independent Ethics Committee or Institutional Review Board | 56 |
| | 9.2 | Ethical Conduct of the Study | 56 |
| | 9.3 | Patient Information and Consent | 56 |
| 10 | Inves | stigator's Obligations | 58 |
| | 10.1 | Confidentiality | 58 |
| | 10.2 | Financial Disclosure and Obligations | 58 |
| | 10.3 | Investigator Documentation | 58 |
| | 10.4 | Study Conduct | 59 |
| | | Adherence to Protocol | |
| | 10.6 | Adverse Events and Study Report Requirements | 59 |
| | 10.7 | Investigator's Final Report | 60 |
| | 10.8 | Records Retention | 60 |
| | 10.9 | Publications | 60 |

Study Management 61

11.1 Monitoring ......61

11

| | | narma, Inc<br>BP-19002 | e.<br>? (Version 2.1) | ABP-450<br>13 May 2021 |
|---|---|---|---|---|
| | | 11.1.1 | External Data Monitoring Committee | 61 |
| | | 11.1.2 | Monitoring of the Study | 61 |
| | | 11.1.3 | Inspection of Records | 61 |
| | 11.2 | Manage | ement of Protocol Amendments and Deviations | 62 |
| | | 11.2.1 | Modification of the Protocol | 62 |
| | | 11.2.2 | Protocol Deviations | 62 |
| | 11.3 | Study 7 | Termination | 62 |
| | 11.4 | Final R | eport | 63 |
| 12 | Refe | rences | | 64 |
| 13 | | | 66 | |
| | 13.2 | TWSTI | RS Scale | 70 |
| | 13.4 | PGI-C | Scale | 76 |
| | 13.5 | | CGI-C Scales | 76 |
| | 13.6 | Dyspha | ngia Severity Scale | |
| | | • • | S Scale | |
| | | | List of Tables | |

Aeon Biopharma, Inc.

Protocol: ABP-19002 (Version 2.1)

ABP-450

13 May 2021

### **Protocol Synopsis**

**Protocol Number:** ABP-19002

**Title:** An Open-Label, Multicenter Study to Evaluate the Safety and

Efficacy of Repeat Intramuscular ABP-450 (prabotulinumtoxinA)

Injection for the Treatment of Cervical Dystonia

**Sponsor:** Aeon Biopharma, Inc.

Study Phase: 2/3

**Study Sites:** Approximate total: 71

United States: 42

**Indication:** Cervical dystonia

Rationale: Cervical dystonia (spasmodic torticollis) is the most common form of

focal dystonia, affecting the neck and shoulder muscles. Cervical dystonia is characterized by abnormal head and neck posture with involuntary head and neck movements. It is often associated with

neck and shoulder pain.

Botulinum toxin A is considered first-line therapy for cervical dystonia, helping to improve pain, posture, and disability. ABP-450 (prabotulinumtoxinA) is a toxin produced by *Clostridium botulinum*. It blocks neuromuscular transmission by binding to acceptor sites on motor nerve terminals, entering the nerve terminals, and inhibiting the release of acetylcholine. Blocking the release of acetylcholine plays a role in relaxing muscles by reducing muscle activity.



ABP-19000 is an ongoing Phase 2, randomized, double-blind, multicenter, placebo-controlled study to evaluate the safety and effectiveness of intramuscular ABP-450 injection for the treatment of cervical dystonia.

ABP-19002 is an open-label extension (OLE) study, wherein eligible patients from ABP-19000 studies, irrespective of treatment allocation, will have the option to continue treatment with ABP-450.

The ABP-19002 study will help to evaluate safety and efficacy of repeat dosing of ABP-450 for the long-term treatment of cervical dystonia.

Objectives:

#### Primary Objective

 To evaluate the safety of repeat intramuscular injections of ABP-450 (150-350 units per dose) in the treatment of cervical dystonia

#### Secondary Objective

• To evaluate the efficacy of repeat intramuscular injections of ABP-450 (150-350 units per dose) in the treatment of cervical dystonia

**Estimands:** 

For all estimands, the target population is patients diagnosed with cervical dystonia. Patients are expected to:

- Have not had previous treatment with BOTOX® within the last 8 weeks
- Have not had previous treatment with ABP-450 within the last 8 weeks
- Be receiving stable doses of treatment for focal dystonia treatment (eg, anticholinergics and benzodiazepines)
- Meet other inclusion/exclusion criteria

**Primary Estimand** 



Secondary Estimands

These are the hypothetical estimands regarding alternative prohibited medications (eg, BOTOX®), assuming (treatment policy) no change in background treatment and administration of treatment within the 150- to 350-unit dose range:



**Study Population:** 

#### **Inclusion Criteria**

Each patient must meet all of the following criteria to be enrolled in this OLE study:

1. Qualified for and had their initial dose of study drug in the ABP-19000

- 2. Provided written informed consent to participate in the study.
- 3. Were a male or female patient between 18 and 75 years of age (inclusive) when they entered the ABP-19000 studies.



6. Stated willingness to comply with all study procedures, including attendance at the study center for all study visits as scheduled and have technological capabilities to have tele visits with video capabilities

#### **Exclusion Criteria**

Patients who meet any of the following criteria will be excluded from this OLE study:



8. Participated in another interventional study during participation in this study.

ABP-450 13 May 2021

Aeon Biopharma, Inc. Protocol: ABP-19002 (Version 2.1)

- 9. Were a pregnant or lactating female, or female of child-bearing potential not willing to use an acceptable method of contraception (ie, intrauterine device, barrier methods with spermicide, or abstinence).
- 10. Would not benefit from treatment with ABP-450 for their cervical dystonia, in the investigator's opinion.
- 11. Viral or other active infection or any medical condition that, in the opinion of the investigator, classifies the patient as unsuitable for participation in the study or patients who do not seem to be in good general health at the time of Screening, and prior to any investigational study drug administration.

Note: Patients will not routinely be tested for COVID-19 during the study. Patients presenting with fever or who are symptomatic for COVID-19 should be treated through their general practitioner.

**Study Design:** 

This is an open-label, Phase 2/3, multicenter, 52-week study of ABP-450 purified neurotoxin complex for the treatment of cervical dystonia. The study population will consist of all patients who had their initial dose of study drug in the ABP-19000 studies, irrespective of treatment allocation, and who consented to being treated for cervical dystonia with ABP-450 in the ABP-19002 OLE study

At the investigator's discretion and with the patient's consent, patients will enter the OLE study at Week 8 (Week 8 will be Day 0 "rollover" for the OLE study) with the opportunity to either maintain the original Phase 2 dose or modify the dose. If there is no efficacy (or loss of efficacy) between 6 and 20 weeks in the ABP-19000 study, then patients can roll over to the OLE study at a dose determined per the investigator's discretion.

**Estimated Study** 

**Safety Assessments:** 

**Duration:** 

| 13 Way 2021 | |
|---|---|
| This OLE study will evaluate the safety and efficacy of repeat | |
| injections of ABP-450 for the long-term treatment of cervical | |
| dystonia. | |
| Deticate will be fellowed on for 52 weeks often they enter the | |
| Patients will be followed up for 52 weeks after they enter the | |
| ABP-19002 OLE study. | |
| Safety will be evaluated by frequency, severity, and duration of an | <b>1</b> 1/ |
| adverse reactions. Adverse events will be assessed at each office | /1S1 |
| and telephone contact. | |
| | 1 |
| | • |
| | _ |

Study Drug, Dosage, and Route of Administration:

Investigational study drug is *Clostridium botulinum* toxin type A. Each vial will contain 100 units of lyophilized ABP-450.

All study patients, regardless of dose group and including placebo patients, will be administered between 150 and 350 units of ABP-450, based on the investigator's discretion and clinical judgment.

The dose should be divided among the affected muscles (see table below). Dosing in initial sessions should be tailored to the individual patient based on the patient's head and neck position, localization of pain, muscle hypertrophy, patient response, and adverse event history.



| Sample Size: | All eligible patients who had their initial dose of study drug in the ABP-19000 studies, irrespective of treatment allocation, and consented to being treated with ABP-450 can be enrolled in this OLE (ie, ABP-19002) study. |
|---|---|
| Statistical Methods: | The proportion of patients with treatment-related SAEs up to Week 52 will be summarized for the Safety Analysis Set with Retreatment. |



Version and Date of Protocol:

Version 2.0 dated 03 December 2020

# **List of Abbreviations**

| Abbreviation | Definition |
|---|---|
| ABP-450 | prabotulinumtoxinA/Jeuveau (prabotulinumtoxinA-xvfs) |
| AE | adverse event |
| $\mathrm{BOTOX}^{\circledR}$ | onabotulinumtoxinA |
| CFR | Code of Federal Regulations |
| CGI-C | Clinical Global Impression of Change |
| CSR | clinical study report |
| C-SSRS | Columbia-Suicide Severity Rating Scale |
| ECG | electrocardiogram |
| eCRF | electronic case report form |
| EMG | electromyographic |
| EOS | end of study |
| FDA | United States Food and Drug Administration |
| FEV <sub>1</sub> | forced expiratory volume in 1 second |
| FVC | forced vital capacity |
| GCP | Good Clinical Practice |
| HbA1c | hemoglobin A1c |
| ICF | informed consent form |
| ICH | International Council for Harmonisation of Technical<br>Requirements for Pharmaceuticals for Human Use |
| IEC | independent ethics committee |
| IRB | institutional review board |

| Abbreviation | Definition |
|--------------|----------------------------------------------------|
| MedDRA | Medical Dictionary for Regulatory Activities |
| mFAS | Modified Full Analysis Set |
| OLE | open-label extension |
| PGI-C | Patient Global Impression of Change |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SAS | Safety Analysis Set |
| SASR | Safety Analysis Set with Retreatment |
| SUSAR | suspected unexpected serious adverse reaction |
| TWSTRS | Toronto Western Spasmodic Torticollis Rating Scale |

#### 1 Introduction

Cervical dystonia (spasmodic torticollis) is the most common form of focal dystonia, affecting the neck and shoulder muscles (Defazio 2004, Mittal 2019). Cervical dystonia is characterized by abnormal head and neck posture with involuntary head and neck movements. It is often associated with neck and shoulder pain.

Botulinum toxin A is considered first-line therapy for cervical dystonia, helping to improve pain, posture, and disability (Comella 2011, Simpson 2016, Mittal 2019). ABP-450 (prabotulinumtoxinA) is a toxin produced by *Clostridium botulinum*. It blocks neuromuscular transmission by binding to acceptor sites on motor nerve terminals, entering the nerve terminals, and inhibiting the release of acetylcholine. Blocking the release of acetylcholine plays a role in relaxing muscles by reducing muscle activity.

| PrabotulinumtoxinA was evaluated in multiple non-clinical safety and toxicological tests to determine the pharmacologic and safety profile of the product in complying with |
|---|
| International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) guidelines/requirements for biologic products. |
| <u>-</u> |



| Aeon Biopharma, Inc. | ABP-450 |
|---|---|
| Protocol: ABP-19002 (Version 2.1) | 13 May 2021 |
| PrabotulinumtoxinA has also been found to be non-inferior to BOTOX moderate to severe glabellar lines in adult patients and upper limb spass stroke (Nam 2015, Rzany 2019). The doses of ABP-450 used in the Philimb spasticity were similar to the doses of BOTOX® used (no signific seen between the 2 groups) (Nam 2015). | sticity in patients with hase 3 study for upper |
| ABP-19000 is an ongoing, Phase 2, randomized, double-blind, multice | enter, |
| placebo-controlled study to evaluate the safety and effectiveness of int | ramuscular ABP-450 |

injection for the treatment of cervical dystonia. ABP-19002 is the open-label extension (OLE) study, wherein eligible patients from ABP-19000 studies, irrespective of treatment allocation, will have the option to continue treatment with ABP-450. The ABP-19002 study will help to evaluate safety and efficacy of repeat dosing of ABP-450 for the long-term treatment of cervical dystonia.

Clostridium botulinum toxins have become the standard of care for the treatment of patients with cervical dystonia, but also have significant risks associated with their use in these patients. The labels of marketed products carry prominent warnings concerning their side effects, such as dysphagia and even death, if they are not carefully administered and the patients are not monitored while under treatment. Even so, the benefit for all these products is greater than the potential risk.

Clinical development of drugs has been impacted by the ongoing COVID-19 pandemic. The current study aims to implement several adjustments or mitigations to allow the study to continue despite pandemic-related disruption. To prioritize patient and site staff safety,

several planned office visits have been converted to tele visits to allow the required data collection to meet the study objectives.

#### 2 Study Objectives and Estimands

#### 2.1 Study Objectives

### 2.1.1 Primary Objective

• To evaluate the safety of repeat intramuscular injections of ABP-450 (150-350 units per dose) in the treatment of cervical dystonia

#### 2.1.2 Secondary Objective

• To evaluate the efficacy of repeat intramuscular injections of ABP-450 (150-350 units per dose) in the treatment of cervical dystonia

### 2.2 Study Estimands

#### 2.2.1 Target Population

For all estimands, the target population is patients diagnosed with cervical dystonia. Patients are expected to:

- Have not had previous treatment with BOTOX® within the last 8 weeks
- Have not had previous treatment with ABP-450 within the last 8 weeks
- Be receiving stable doses of treatment for focal dystonia treatment (eg, anticholinergics and benzodiazepines)
- Meet other inclusion/exclusion criteria

# 2.2.2 Primary Estimand

| The | primary | estimand | of the | study | will | be: |
|-----|---------|----------|--------|-------|------|-----|
|-----|---------|----------|--------|-------|------|-----|



## 2.2.3 Secondary Estimands

These are the hypothetical estimands regarding alternative prohibited medications (eg, BOTOX®), assuming (treatment policy) no change in background treatment and administration of treatment within the 150- to 350-unit dose range:



# 3 Investigational Plan

# 3.1 Study Design

| This is an open-label, Phase 2/3, multicenter, 52-week study of ABP-450 purified neurotoxin complex for the treatment of cervical dystonia. The study population in the ABP-19002 OLE study will consist of all patients who had their initial dose of study drug in the ABP-19000 studies, irrespective of treatment allocation, who consented to being treated for cervical dystonia with ABP-450, |
|---|
| At the investigator's discretion and with the patient's consent, patients will enter the OLE study at Week 8 (Week 8 will be Day 0 "rollover" for the OLE study) with the opportunity to either maintain the original Phase 2 dose or modify the dose. If there is no efficacy (or loss of efficacy) between 6 and 20 weeks in the ABP-19000 study, then patients can roll over to the OLE study at a dose determined per the investigator's discretion. |
| During this OLE study, patients will receive any dose between 150 and 350 units of ABP-450, based on the investigator's discretion. There will be no additional retreatments after Week 48. |
| This OLE study will evaluate the safety and efficacy of repeat injections of ABP-450 for the long-term treatment of cervical dystonia. 3.1.1 Rationale of Study Design |
| 5.1.1 Kationale of Study Design |

### 3.1.2 Conduct of the Study During the COVID-19 Pandemic

Coronavirus Disease 2019 (COVID-19) is a viral illness caused by the severe acute respiratory syndrome-related coronavirus 2 (SARS-CoV-2) and has impacted most of the countries across the globe. It was declared as a global public health emergency by the World Health Organization on 30 January 2020. This pandemic is recognized to have impacted the conduct of clinical trials of medical products in various ways.

The safety and well-being of patients and site staff is of paramount importance during the COVID-19 pandemic. Measures will be implemented during the study to reduce the chance that study drug will be administered to patients who are infected with SARS-CoV-2.

Testing for COVID-19 will be performed as required by the individual sites in case deemed necessary by the PI as per institutional standards. If a patient tests positive, study visits related to retreatment will be delayed until patient recovers. The investigator will provide the patients with guidance of further clinical care for their SARS-CoV-2 infection. If the result is indeterminate, the PCR testing may need to be repeated as per institutional standards.

Other potential measures will be taken to assure the safety and welfare of patients, maintaining compliance with GCP, and minimizing risks to trial integrity during the COVID-19 pandemic, such as tele visits. Any other potential measures or changes will be handled according to the regulations.

Any events of COVID-19, including asymptomatic and symptomatic SARS-CoV-2 infection (i.e., COVID-19), are to be reported as AEs per Section 6.2.1.

All the measures taken in relation to COVID-19 will be reported to the regulatory authorities as appropriate.

## 4 Patient Selection and Withdrawal Criteria

# 4.1 Selection of Study Population

| irrespe | ctiv | studies, see of treatment allocation, and who consented to being treated for cervical dystonia 450 will be eligible to enroll in this OLE study The study will be conducted at approximately 42 sites in the United States Patients will be administered investigational |
|---|---|---|
| study d | lrug | g only if they meet all of the inclusion criteria and none of the exclusion criteria. |
| | | ho fail their initial Screening will be allowed to present for rescreening once, if in advance by the medical monitor (see Section 4.1.3). |
| 4.1.1 | In | clusion Criteria |
| Each p | atie | nt must meet all of the following criteria to be enrolled in this OLE study: |
| | 1. | Qualified for and had their initial dose of study drug in the ABP-19000 |
| | 2 | |
| | 2. | Provided written informed consent to being treated for cervical dystonia with ABP-450. |
| | 3. | Were a male or female patient between 18 and 75 years of age (inclusive) when they entered the ABP-19000 studies. |

#### 4.1.2 Exclusion Criteria

Patients who meet any of the following criteria will be excluded from this OLE study:



- 8. Participated in another interventional study during participation in this study.
- 9. Were a pregnant or lactating female, or female of child-bearing potential not willing to use an acceptable method of contraception (ie, intrauterine device, barrier methods with spermicide, or abstinence).
- 10. Would not benefit from treatment with ABP-450 for their cervical dystonia, in the investigator's opinion.
- 11. Viral or other active infection or any medical condition that, in the opinion of the investigator, classifies the patient as unsuitable for participation in the study or patients who do not seem to be in good general health at the time of Day 0 "rollover", and prior to any investigational study drug administration.

Note: Patients will not routinely be tested for COVID-19 during the study. Patients presenting with fever or who are symptomatic for COVID-19 should be treated through their general practitioner.

### 4.1.3 Rescreening

A screen failure is a patient who has given informed consent and failed to meet all of the inclusion criteria and/or met at least one of the exclusion criteria and has not been randomized (eg, due to a viral or other active infection, or repeat laboratory test result outside of reference range). Patients who fail their initial Screening will be allowed to present for rescreening once, if approved in advance by the medical monitor. Rescreen requests must be discussed with the medical monitor prior to rescreening the patient, including what has changed about the patient's medical status.

Patients who present for rescreening will be assigned a new Screening number. The investigator or designee will record rescreening data on the source document and the appropriate eCRF. Details for rescreening procedures will be provided in the IRT manual.

### 4.2 Withdrawal of Patients from the Study

Patients will be followed up for 52 weeks after they enter the ABP-19002 OLE study.

#### 4.2.1 Reasons for Withdrawal/Discontinuation

Patients may withdraw from the study at any time and for any reason without prejudice to their future medical care by the investigator or at the study site. Every effort should be made to keep patients in the study. The reasons for patients not completing the study will be recorded. A patient may be withdrawn from the study for any of the following reasons:





8. The patient withdraws consent.

The investigator will also withdraw a patient if Aeon Biopharma, Inc. terminates the study. Upon occurrence of a serious or intolerable AE, the investigator will confer with the sponsor. If a patient is discontinued because of an AE, the event will be followed until it is resolved. Any patient may withdraw his or her consent at any time.

#### 4.2.2 Handling of Withdrawals

Patients are free to withdraw from the study or study treatment at any time at their request. Patient participation in the study may be stopped at any time at the discretion of the investigator or at the request of the sponsor.



It is vital to obtain follow-up data on any patient withdrawn because of an AE or SAE. In every case, efforts must be made to undertake protocol-specified safety follow-up procedures. All data collected from all patients, including early withdrawals and early discontinuations of treatment, will be used in the reporting and analysis of the study.

## 4.2.3 Replacements

Patients who discontinue prematurely from the study will not be replaced.

## **5 Study Treatments**

# 5.1 Method of Assigning Patients to Treatment Group

| Patients who meet all eligibility criteria will continue the current OLE study with the randomization code assigned by an interactive response technology system in the ABP-19000 studies as their study number. All eligible patients who had their initial dose of study drug in the ABP-19000 studies, irrespective of treatment allocation, and who consented to being treated for cervical dystonia, |
|---|
| receive ABP-450 in an unblinded fashion. |
| 5.2 Treatment Administered |
| Investigational study drug is a <i>Clostridium botulinum</i> toxin type A. Each vial will contain 100 units of lyophilized ABP-450. |
| The ABP-450 dose to be administered to patients in the ABP-19002 OLE study will range between 150 and 350 units. Patients will be enrolled in the ABP-19002 OLE study with the opportunity to either maintain or modify the dose at the investigator's discretion. As the blind will not be broken, the placebo patients (who were entered into one of the dose groups in the ABP-19000 studies) can be administered any dose between 150 and 350 units of ABP-450, based on the investigator's discretion and clinical judgment. |


| 5.3 | <b>Identity of Investigational Product</b> |
|---|---|
| ABP- | 450 is a lyophilized powder packed in vials, each containing 100 units. |
| 5.4 | Management of Clinical Supplies |
| 5.4.1 | Investigational Study Drug Packaging and Storage |

# 5.4.2 Test Article Accountability

The investigator will maintain accurate records of receipt of test article, including dates of receipt. In addition, accurate records will be kept regarding when and how much test article is dispensed and used by each patient in the study. Reasons for departure from the expected dispensing regimen must also be recorded. At the completion of the study, to satisfy

regulatory requirements regarding drug accountability, investigational study drug will be reconciled and retained or destroyed according to applicable regulations.

#### **5.4.3** Other Supplies



#### 5.5 Overdose Management

An overdose is any dose of investigational study drug given to a patient or taken by a patient that exceeds the dose described in the protocol. Any overdose, with or without associated AEs, must be promptly reported to the symptoms do not need to be recorded as AEs; in case of any AEs associated with the overdose, these should be reported on relevant AE/SAE sections of the eCRF.

#### **5.5.1** Treatment of Overdose

Treatment of suspected overdose of investigational study drug should include investigational study drug discontinuation and implementation of appropriate supportive measures.

#### 5.6 Blinding

This is an OLE study. All eligible patients from the ABP-19002 studies will receive ABP-450 in an unblinded fashion. As the blind will not be broken, the placebo patients (who were entered into one of the dose groups in the ABP-19000 studies) can be administered any dose between 150 and 350 units of ABP-450, based on the investigator's discretion.

# **5.6.1** Breaking the Blind

Not applicable, as this is an OLE study.

# 5.7 Treatment Compliance

Patient compliance will be determined by capturing the precise dose administered and the time and date of dosing in the source document and the dosage administration eCRF. Delays in dosing and the reason for any delay in dosing are to be recorded on the dosage administration eCRF.

# 5.8 Prior and Concomitant Therapy

Use of all concomitant medications will be recorded in the patient's eCRF. The minimum requirement is that drug name, dose, route of administration, reason for taking, and dates of administration are to be recorded. This will include all prescription drugs, herbal products, vitamins, minerals, and over-the-counter medications. Any changes in concomitant medications also will be recorded in the patient's eCRF.

Any concomitant medication deemed necessary for the welfare of the patient during the study may be given at the discretion of the investigator. However, it is the responsibility of the investigator to ensure that details regarding the medication are recorded in full in the eCRF.

# **6** Study Assessments and Procedures

Before performing any study procedures, all potential patients will sign an informed consent form (ICF) for this OLE study. Patients will have the opportunity to have any questions answered before they sign the ICF. The investigator must address all questions raised by the patient. The investigator will also sign the ICF.

#### 6.1 Study Visits

Patients will be followed up for 52 weeks after they enter the ABP 19002 OLE study.





| • | |
|---|---|
| • | |
| • | |
| • | |
| Safe | ty Assessments |
| | e evaluated by frequency, severity, and duration of any adverse reactions.<br>nts will be assessed at each office visit and telephone contact. |

#### **6.2.1** Adverse Events

#### **6.2.1.1** Definitions of Adverse Events

The investigator is responsible for reporting all AEs that are observed or reported during the study, regardless of their relationship to investigational study drug. The investigator will query the patient for changes since last visit and ask about the patient's ability to swallow.

An AE is defined as any untoward medical occurrence in a patient enrolled into this study regardless of its causal relationship to investigational study drug. Patients will be instructed to contact the investigator at any time after enrollment if any symptoms develop.

A treatment-emergent AE is defined as any event not present before exposure to investigational study drug or any event already present that worsens in either intensity or frequency after exposure to investigational study drug.

#### **6.2.1.2** Serious Adverse Events

An SAE is defined as any event that

- results in death
- is immediately life-threatening
- requires inpatient hospitalization or prolongation of existing hospitalization
- results in persistent or significant disability/incapacity
- is a congenital anomaly/birth defect



# **6.2.1.3** Eliciting and Documenting Adverse Events

Adverse events will be assessed from the time the patient signs the ICF until exit from the study (ie, 52 weeks or end of treatment [ET] after Day 0 "rollover").

Serious AEs that occur more than 56 days (ie, 8 weeks) after the last dose of investigational study drug and the patient has exited the study need not be reported unless the investigator considers them related to investigational study drug.

At every study visit, patients will be asked a standard non-leading question to elicit any medically related changes in their well-being. They will also be asked if they have been hospitalized, had any accidents, used any new medications, or changed concomitant medication regimens (both prescription and over-the-counter medications).

In addition to patient observations, AEs identified from any study data (eg, laboratory values, physical examination findings, changes in 12-lead ECG results) or identified from review of other documents that are relevant to patient safety will be documented on the AE page in the eCRF.

#### **6.2.1.4** Reporting Adverse Events

All AEs reported or observed during the study will be recorded on the AE page in the eCRF. Information to be collected includes the following:

- Drug treatment
- Dose
- Event term
- Time of onset
- Investigator-specified assessment of severity and relationship to investigational study drug
- Time of resolution of the event
- Seriousness
- Any required treatment or evaluations
- Outcome

Adverse events resulting from concurrent illnesses, reactions to concurrent illnesses, reactions to concurrent medications, or progression of disease states must also be reported. All AEs will be followed to adequate resolution. The Medical Dictionary for Regulatory Activities (MedDRA) will be used to code all AEs.

Any medical condition that is present at the time that the patient is screened but does not deteriorate should not be reported as an AE. However, if it deteriorates at any time after Screening Visit, it should be recorded as an AE.

#### **6.2.1.5** Reporting Serious Adverse Events



Sponsor or its designee is responsible for reporting relevant SAEs to the competent authority, other applicable regulatory authorities, and participating investigators, in accordance with the ICH guidelines and/or local regulatory requirements.

The sponsor is responsible for reporting unexpected fatal or life-threatening events associated with the use of investigational study drug (expedited reports) to the regulatory agencies and competent authorities by telephone or fax within 7 calendar days after being notified of the event. The sponsor should report other relevant SAEs associated with the use of investigational study drug to the appropriate competent authorities (according to local guidelines), investigators, and the institutional review board (IRB) by a written safety report within 15 calendar days of notification.

# 6.2.1.6 Suspected Unexpected Serious Adverse Reactions and Non-Serious Adverse Events of Special Interest

The sponsor will promptly evaluate all suspected unexpected serious adverse reactions (SUSARs) and non-serious AEs of special interest against cumulative investigational study drug experience to identify and expeditiously communicate possible new safety findings to investigators, IRBs/independent ethics committees (IECs), and applicable health authorities based on applicable legislation.



#### **6.2.1.7** Assessment of Severity

The severity, or intensity, of an AE refers to the extent to which an AE affects the patient's daily activities. The intensity of the AE will be rated as mild, moderate, or severe using the following criteria:

Mild: An event usually transient in nature and generally not interfering with normal

activities.

Moderate: An AE that is sufficiently discomforting to interfere with normal activities.

Severe: An AE that is incapacitating and prevents normal activities.

Changes in the severity of an AE should be documented to allow an assessment of the duration of the event at each level of intensity to be performed. AEs characterized as intermittent do not require documentation of onset and duration of each episode.

#### **6.2.1.8** Assessment of Causality

The investigator's assessment of an AE's relationship to investigational study drug is part of the documentation process, but it is not a factor in determining what is or is not reported in the study. If there is any doubt as to whether a clinical observation is an AE, the event should be reported.

The relationship or association of the test article in causing or contributing to the AE will be characterized using the following classification and criteria:

<u>Unrelated</u>: This relationship suggests that there is no association between investigational

study drug and the reported event.

<u>Possible</u>: This relationship suggests that treatment with investigational study drug

caused or contributed to the AE, ie, the event follows a reasonable temporal sequence from the time of drug administration or follows a known response pattern to investigational study drug but could also have been produced by

other factors.

<u>Unrelated</u>: This relationship suggests that there is no association between investigational study drug and the reported event.

Probable: This relationship suggests that a reasonable temporal sequence of the event

with drug administration exists and, based upon the known pharmacological action of the drug, known or previously reported adverse reactions to the drug or class of drugs, or judgment based on the investigator's clinical experience, the association of the event with investigational study drug seems likely. The event disappears or decreases on cessation or reduction of the dose of

investigational study drug.

<u>Definite</u>: This relationship suggests that a definite causal relationship exists between

drug administration and the AE, and other conditions (concurrent illness, progression or expression of disease state, or concurrent medication reaction) do not appear to explain the event. The event reappears or worsens if the

investigational study drug is re-administered.

#### **6.2.1.9** Follow-Up of Patients Reporting Adverse Events

All AEs must be reported in detail on the appropriate page in the eCRF and followed to satisfactory resolution, until the investigator deems the event to be chronic or not clinically significant, or until the patient is considered to be stable.

# 6.3 Secondary Efficacy Assessments

#### 6.3.1 TWSTRS Scale

Most studies leading to the approval of currently available botulinum neurotoxins have used the TWSTRS scale as the primary efficacy measure (Fernandez 2013; Espay 2018). The standard TWSTRS is a comprehensive scale that comprises three subsets to assess motor severity, pain, and disability (Comella 2016). The motor severity subscale consists of 10 items, with variable scaling and weighting. It also includes a disability subscale with 7 items, and a pain scale with 3 items. The total score is the sum of each of the subscales.

#### 6.3.2 PGI-C and CGI-C Scales

The PGI-C enables the patient to rate changes in their perception of their general health status over the duration of the assessment via a 7-point scale ranging from "very much improved" to "very much worse" (Fischer 1999). For this study, a 5-point generic PGI-C scale ranging from "much better" to "much worse" was used (FDA 2018). Similarly, the CGI-C is a 7-point scale ranging from "very much improved" to "very much worse" (Guy 1976) based on the physician's perception of the patient's health status. Detailed descriptions of the PGI-C and CGI-C are provided in Appendix 13.4 and Appendix 0, respectively.



#### **6.3.4 C-SSRS**

The C-SSRS was developed by the FDA in 2012 for measuring suicidal ideation and behavior in clinical trials (Posner 2011). The C-SSRS was designed to distinguish the domains of suicidal ideation and suicidal behavior. Four constructs are measured. The first is the severity of ideation (hereafter referred to as the "severity subscale"), which is rated on a 5-point ordinal scale in which 1=wish to be dead, 2=non-specific active suicidal thoughts, 3=suicidal thoughts with methods, 4=suicidal intent, and 5=suicidal intent with plan. The second is the intensity of ideation subscale (hereafter referred to as the "intensity subscale"), which comprises five items, each rated on a 5-point ordinal scale: frequency, duration, controllability, deterrents, and reason for ideation. The third is the "behavior subscale," which is rated on a nominal scale that includes actual, aborted, and interrupted attempts; preparatory behavior; and non-suicidal self-injurious behavior. The fourth is the "lethality subscale," which assesses actual attempts; actual lethality is rated on a 6-point ordinal scale,

and if actual lethality is zero, potential lethality of attempts is rated on a 3-point ordinal scale (Posner 2011). A detailed description is provided in Appendix 13.7.

| 6.3.5 | Dysphagia Score |
|---|---|
| 6.4 | Safety Monitoring Committee |
| | nedical monitor and sponsor will hold monthly reviews of all AEs; consequently, an endent Safety Committee will not be formed for this study. |
| 6.5 | Pregnancy |
| 6.6 | Laboratory Analyses |
| Any a | bnormal laboratory test results |
| | including those that worsen from Day 0 "rollover," felt to be clinically |

| Protocol: ABP-19002 (Version 2.1) | 13 May 2021 |
|---|---|
| significant in the medical and scientific judgment of the investigator are to be real. AEs or SAEs. | ecorded as |
| However, any clinically significant safety assessments that are associated with t disease, unless judged by the investigator to be more severe than expected for the condition, are not to be reported as AEs or SAEs. | , , |
| 6.7 Sample Collections | |
| Site personnel will collect blood samples at the visits specified in Section 6.1. T will be processed at the site and shipped same day to a central laboratory, as spelaboratory manual. | - |

Aeon Biopharma, Inc.

ABP-450

#### 7 Statistical Considerations

This section briefly describes statistical and analytical methods to be used for the study. A statistical analysis plan (SAP) will provide details of the statistical methods and definitions for the analysis of efficacy and safety data. To preserve the integrity of the statistical analysis and study conclusions, the SAP will be finalized before database lock.

#### 7.1 Estimands

# 7.2 Sample Size Calculations

All eligible patients who had their initial dose of study drug in the ABP-19000 studies, irrespective of treatment allocation, and consented to being treated with ABP-450 will be eligible to enroll in this OLE study.

Approximately 60 patients could enroll in this OLE study from the ABP-19000 study,

#### 7.3 Analysis Sets

The following analysis sets will be used in the statistical analyses.

<u>Full Analysis Set (FAS)</u>: The FAS will consist of all patients who received investigational study drug.

Modified Full Analysis Set (mFAS): The mFAS will consist of all patients in the FAS but will exclude data points

<u>Per-Protocol Analysis Set</u>: The Per-Protocol Analysis Set will consist of all patients in the FAS who received ABP-450 within the study dose range of 150 to 350 units but will exclude all patients who had significant protocol violations or do not receive more than one treatment of ABP-450 within the OLE study.

<u>Safety Analysis Set (SAS)</u>: The SAS will consist of all patients who received investigational study drug.

| | ABP-450 |
|----|----------|
| 13 | May 2021 |

Aeon Biopharma, Inc. Protocol: ABP-19002 (Version 2.1)

<u>Safety Analysis Set with Retreatment (SASR)</u>: The SASR will consist of all patients in the SAS but will exclude patients who do not receive more than one treatment of ABP-450 within the OLE study.

# 7.4 Description of Subgroups to be Analyzed

No subgroup analyses are planned.

#### 7.5 Statistical Analysis Methodology

Variables will generally be summarized using number of observations, mean, standard deviation, median, minimum, maximum, and missing data (for continuous variables) and using frequencies, percentages, and missing data (for categorical variables). Data will be listed in data listings.

Details of the statistical analyses, methods, and data conventions will be described in the SAP.

### 7.5.1 Analysis of Primary Estimand

The proportion of patients with treatment-related SAEs up to Week 52 will be summarized for the SASR.

# 7.5.2 Analysis of Secondary Estimands The analysis of the first secondary efficacy estimand is based on a regression model with change

# 7.5.3 Other Analyses

Summary statistical analyses will be provided for demographics, background characteristics, medical history, and physical examination.

# 7.5.4 Interim Analyses

No interim analyses are planned.

#### 8 Data Quality Assurance

The sponsor or its designee will perform the quality assurance and quality control activities of this OLE study, including regular monitoring visits to study sites and meeting with site personnel. However, the investigator generating the data will be responsible for the accuracy, completeness, and reliability of the study data presented to the sponsor.

#### 8.1 Data Management

As part of the responsibilities assumed by participating in the study, the investigator agrees to maintain adequate case histories for the patients treated as part of the research under this protocol. The investigator agrees to maintain accurate eCRFs and source documentation as part of the case histories. These source documents may include laboratory reports

All eCRF information is to be filled in. If an item is not available or is not applicable, this fact should be indicated. Blank spaces should not be present unless otherwise directed. A correction to source documentation should be made by striking through the incorrect entry with a single line and the corrected information should be entered adjacent to the deleted item. The correction must be initialed and dated by the person making the correction.

Investigative site personnel will enter patient data into an electronic data capture system. The analysis data sets will be a combination of these data and data from other sources (eg, laboratory data).

Clinical data management will be performed in accordance with applicable Aeon Biopharma, Inc. standards and data cleaning procedures to ensure the integrity of the data (eg, removing errors and inconsistencies in the data). Adverse event terms will be coded using MedDRA, an internal validated medical dictionary, and concomitant medications will be coded using the World Health Organization Drug Dictionary.



#### 9 Ethics

#### 9.1 Independent Ethics Committee or Institutional Review Board

Federal regulations and the ICH guidelines require that approval be obtained from an IRB/IEC before participation of human patients in research studies. Before study onset, the protocol, informed consent, advertisements to be used for the recruitment of study patients, and any other written information regarding this study to be provided to the patient must be approved by the IRB/IEC. Documentation of all IRB/IEC approvals and of the IRB/IEC compliance with ICH guideline E6 (R2): Good Clinical Practice (GCP) will be maintained by the site and will be available for review by the sponsor or its designee.

All IRB/IEC approvals should be signed by the IRB/IEC chairman or designee and must identify the IRB/IEC name and address, the clinical protocol by title or protocol number or both, and the date of approval or a favorable opinion was granted.

The investigator is responsible for providing written summaries of the progress and status of the study at intervals not exceeding 1 year or otherwise specified by the IRB/IEC. The investigator must promptly supply the sponsor or its designee, the IRB/IEC, and where applicable, the institution, with written reports on any changes significantly affecting the conduct of the study or increasing the risk to patients.

# 9.2 Ethical Conduct of the Study

The study will be performed in accordance with the ethical principles that have their origin in the Declaration of Helsinki, ICH GCP, the protocol, and all applicable regulations.

#### 9.3 Patient Information and Consent

A written informed consent in compliance with United States Title 21 Code of Federal Regulations (CFR) Part 50 shall be obtained from each patient before entering the study or performing any study procedure. An informed consent template may be provided by the sponsor to investigative sites. If any institution-specific modifications to study-related procedures are proposed or made by the site, the consent should be reviewed by the sponsor or its designee or both before IRB/IEC submission. Once reviewed, the consent will be submitted by the investigator to his or her IRB/IEC for review and approval before the start of the study. If the ICF is revised during the course of the study, all active participating patients must sign the revised form.

Before recruitment and enrollment, each prospective patient will be given a full explanation of the study and be allowed to read the approved ICF. Once the investigator is assured that

the patient understands the implications of participating in the study, the patient will be asked to give consent to participate in the study by signing the ICF.

The investigator shall retain the signed original ICF(s) and give a copy of the signed original form to the patient.

#### 10 Investigator's Obligations

The following administrative items are meant to guide the investigator in the conduct of the study but may be subject to change based on industry and government standard operating procedures, working practice documents, or guidelines. Administrative changes will be reported to the IRB/IEC but will not result in protocol amendments.

#### 10.1 Confidentiality

All laboratory specimens, evaluation forms, reports, and other records will be identified in a manner designed to maintain patient confidentiality. All records will be kept in a secure storage area with limited access. Clinical information will not be released without the written permission of the patient, except as necessary for monitoring and auditing by the sponsor, its designee, the FDA, or the IRB/IEC.

The investigator and all employees and coworkers involved with this study may not disclose or use for any purpose other than performance of the study any data, record, or other unpublished, confidential information disclosed to those individuals for the purpose of the study. Prior written agreement from the sponsor or its designee must be obtained for the disclosure of any said confidential information to other parties.

#### 10.2 Financial Disclosure and Obligations

Investigators are required to provide financial disclosure information to allow the sponsor to submit the complete and accurate certification or disclosure statements required under 21 CFR 54. In addition, the investigator must provide to the sponsor a commitment to promptly update this information if any relevant changes occur during the course of the investigation and for 1 year following the completion of the study.

Neither the sponsor is financially responsible for further testing or treatment of any medical condition that may be detected during the Screening process. In addition, in the absence of specific arrangements, neither the sponsor is financially responsible for further treatment of the patient's disease.

# 10.3 Investigator Documentation

Prior to beginning the study, the investigator will be asked to comply with ICH E6 (R2) 8.2 and Title 21 of the CFR by providing the following essential documents, including but not limited to:

IRB/IEC approval

- Original investigator-signed investigator agreement page of the protocol
- Form FDA 1572, fully executed, and all updates on a new fully executed Form FDA 1572 (applicable to study sites in the United States only)
- Curriculum vitae for the investigator and each subinvestigator listed on Form FDA 1572 (applicable to study sites in the United States only)
- Financial disclosure information to allow the sponsor to submit complete and accurate certification or disclosure statements required under 21 CFR 54. In addition, the investigators must provide to the sponsor a commitment to promptly update this information if any relevant changes occur during the course of the investigation and for 1 year after the completion of the study
- IRB/IEC-approved informed consent, samples of site advertisements for recruitment for this study, and any other written information regarding this study that is to be provided to the patient
- Laboratory certifications and normal ranges for any local laboratories used by the site, in accordance with 42 CFR 493

#### 10.4 Study Conduct

The investigator agrees that the study will be conducted according to the principles of ICH E6 (R2). The investigator will conduct all aspects of this study in accordance with all national, state, and local laws or regulations. Study information from this protocol will be posted on publicly available clinical trial registers before enrollment of patients begins.

#### 10.5 Adherence to Protocol

The investigator agrees to conduct the study as outlined in this protocol in accordance with ICH E6 (R2) and all applicable guidelines and regulations.

# 10.6 Adverse Events and Study Report Requirements

By participating in this study, the investigator agrees to submit reports of SAEs to the sponsor and/or IRB/IEC according to the timeline and method outlined in the protocol. In addition, the investigator agrees to submit annual reports to the study site IRB/IEC as appropriate.

#### 10.7 Investigator's Final Report

Upon completion of the study, the investigator, where applicable, should inform the institution; the investigator/institution should provide the IRB/IEC with a summary of the study's outcome and the sponsor and regulatory authorities with any reports required.

#### 10.8 Records Retention

Essential documents should be retained until at least 2 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or at least 2 years have elapsed since the formal discontinuation of clinical development of the investigational study drug. These documents should be retained for a longer period, however, if required by the applicable regulatory requirements or by an agreement with the sponsor. It is the responsibility of the sponsor to inform the investigator/institution as to when these documents no longer need to be retained.

#### 10.9 Publications

After completion of the study, the data may be considered for reporting at a scientific meeting or for publication in a scientific journal. In these cases, the sponsor will be responsible for these activities and will work with the investigators to determine how the manuscript is written and edited, the number and order of authors, the publication to which it will be submitted, and other related issues. The sponsor has final approval authority over all such issues.

Data are the property of the sponsor and cannot be published without prior authorization from the sponsor, but data and publication thereof will not be unduly withheld.

#### 11 Study Management

The administrative structure will include a scientific steering committee and event adjudication committee.

The scientific steering committee, composed of key opinion leaders expert in the treatment of patients with cervical dystonia, will consult with the sponsor on the design of the study protocol, review the data, and analyze the data incorporated into the final study report.

# 11.1 Monitoring

# 11.1.1 External Data Monitoring Committee

No data monitoring committee is planned for this study.

# 11.1.2 Monitoring of the Study

| The clinical monitor, as a representative of the sponsor, has the obligation to follow the study |
|---|
| closely. |
| 11.1.3 Inspection of Records |
| Investigators and institutions involved in the study will permit study-related monitoring, audits, IRB/IEC review, and regulatory inspections by providing direct access to all study |
| records. |

#### 11.2 Management of Protocol Amendments and Deviations

#### 11.2.1 Modification of the Protocol

Any changes in this research activity, except those necessary to remove an apparent, immediate hazard to the patient, must be reviewed and approved by the sponsor or its designee. Amendments to the protocol must be submitted in writing to the investigator's IRB/IEC for approval before patients can be enrolled into an amended protocol.

#### 11.2.2 Protocol Deviations

| The investigator or designee must document and explain in the patient's source |
|---|
| documentation any deviation from the approved protocol. |

# 11.3 Study Termination

Although Aeon Biopharma, Inc. has every intention of completing the study, Aeon Biopharma, Inc. reserves the right to discontinue the study at any time for clinical or administrative reasons.

The end of the study is defined as the date on which the last patient completes the EOS visit (ie, 52 weeks after Day 0 "rollover"), patient withdrawal (for any reason), or study discontinuation by the sponsor.

# 11.4 Final Report

Whether the study is completed or prematurely terminated, the sponsor will ensure that the clinical study reports (CSRs) are prepared and provided to the regulatory agencies as required by the applicable regulatory requirements. The sponsor will also ensure that the CSRs in marketing applications meet the standards of the ICH guideline E3: Structure and Content of Clinical Study Reports.

Where required by applicable regulatory requirements, an investigator signatory will be identified for the approval of the CSR. The investigator will be provided reasonable access to statistical tables, figures, and relevant reports and will have the opportunity to review the complete study results.

Upon completion of the CSR, the sponsor will provide the investigator with the full summary of the study results. The investigator is encouraged to share the summary results with the study patients, as appropriate. The study results will be posted on publicly available clinical trial registers.

# 12 References



| Protocol: ABP-19002 (Version 2.1) | 13 May 202 |
|-----------------------------------|------------|

Aeon Biopharma, Inc.

ABP-450

# 13 Appendices



Page 66







# 13.2 TWSTRS Scale













# 13.4 PGI-C Scale







# 13.6 Dysphagia Severity Scale



# 13.7 C-SSRS Scale



